CLINICAL TRIAL: NCT06613009
Title: A Phase 1 Multicenter, Open-label Study of IBI3009 in Participants with Unresectable, Metastatic or Extensive-Stage Small Cell Lung Cancer
Brief Title: Study of IBI3009 in Participants with Unresectable, Metastatic or Extensive-Stage Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI3009A101
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IBI3009 (Experimental)
  Interventions: Drug: IBI3009

INTERVENTIONS:
Drug: IBI3009 — Monoclonal Antibody-Camptothecin Derivative Conjugate for Injection (R & D code: IBI3009)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of IBI3009 and to determine the maximum tolerated dose (MTD) and/or the recommended dose for expansion (RDE) of IBI3009.

ELIGIBILITY:
Inclusion Criteria:

1. Participants have the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol;
2. Male or female subjects ≥ 18 years old. For Part 1, age ≥18 years and ≤75 years;
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-1;
4. Minimum life expectancy of ≥ 12 weeks;
5. Adequate organ function confirmed at screening period;
6. Histologically or cytologically confirmed unresectable,metastatic or Extensive-Stage small cell lung cancer (SCLC).

Exclusion Criteria

1. Participating in any other interventional clinical research except observational (non-interventional) study or in the follow-up phase of an interventional study;
2. Has adverse reactions resulting from previous anti-tumor therapies, which have not resolved to Grade 0 or 1 toxicity according to NCI CTCAE v5.0 (except for alopecia, fatigue, pigmentation and other conditions with no safety risk according to investigator's discretion) prior to the first dose of the study drug;
3. Known allergies, hypersensitivity, or intolerance to IBI3009 or its excipients;
4. Undergone major surgery (Craniotomy, thoracotomy or laparotomy, and other surgery according to investigator's discretion, excluding needle biopsy) within 4 weeks prior to the first dose of the study drug, or who are expected to undergo major surgery during the study period, or who have severe unhealed wounds, trauma, ulcers, etc.;
5. Women who are pregnant, have positive results in pregnancy test or are lactating;
6. Not eligible to participate in this study at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Numbers of subjects with adverse events | Up to 3 years
  defined as any untoward medical occurrence, whether or not there is a causal relationship with the study drug, in a clinical study subject from the time informed consent form is signed
Number of subjects with clinically significant changes in physical examination results | Up to 3 years
  Clinically significant abnormal physical examination findings reported by the investigator.
Number of subjects with clinically significant changes in electrocardiogram | Up to 3 years
  Clinically significant abnormal electrocardiogram findings reported by the investigator.
Number of subjects with clinically significant changes in vital signs | Up to 3 years
  Vital signs including body temperature, pulse, respiratory rate, SpO2 and blood pressure
Dose limiting toxicities (DLTs) | Up to 28 days
  Dose limiting toxicities (DLTs) to establish MTD and/or RDE.

SECONDARY OUTCOMES:
area under the curve (AUC) | Up to 3 years
  area under the curve (AUC) of single and multiple doses of IBI3009
maximum concentration (Cmax) | Up to 3 years
  maximum concentration (Cmax) of single and multiple doses of IBI3009
time to maximum concentration (Tmax) | Up to 3 years
  time to maximum concentration (Tmax) of single and multiple doses of IBI3009
clearance (CL) | Up to 3 years
  clearance (CL) of single and multiple doses of IBI3009
apparent volume of distribution (V) | Up to 3 years
  apparent volume of distribution (V) of single and multiple doses of IBI3009
half-life (t1/2) | Up to 3 years
  half-life (t1/2) of IBI3009 to the last administration of IBI3009
anti-drug antibody (ADA) | Up to 3 years
  Incidence and characterization of anti-drug antibody (ADA).
objective response rate (ORR) | Up to 3 years
  objective response rate (ORR) as evaluated per the RECIST v1.1 criteria.
duration of response (DoR) | Up to 3 years
  duration of response (DoR) as evaluated per the RECIST v1.1 criteria.
time to response (TTR) | Up to 3 years
  time to response (TTR) as evaluated per the RECIST v1.1 criteria.
progression free survival (PFS) | Up to 3 years
  as evaluated per the RECIST v1.1 criteria.
overall survival (OS) | Through out the study (an average of 3 years)
  OS is defined as the time from the date of first dose of study drug until the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Austin Hospital, Heidelberg, Victoria
- China (7):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Cancer Hospital of Shandong First Medical University(Shandong Cancer Institute, Shandong Cancer Hospital), Jinan, Shandong
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No